CLINICAL TRIAL: NCT05032482
Title: WeArable Neuromodulation DeVice for the TrEatment of Alzheimer's Disease
Acronym: WAVE-AD
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding purposes
Sponsor: Scion NeuroStim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNS-AD-001
Record Dates: First submitted 2021-08-26; First posted 2021-09-02 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Mild Alzheimer's Disease
Keywords: Open Label Extension; Medical Devices; Non-Invasive Brain Stimulation; Randomized Controlled Trial; Brainstem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The first 24 weeks will be the randomized controlled portion of the study; the remaining 24 weeks will be an open label extension.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (3):
- Investigational Treatment 1 (Other): Investigational treatment mode (stimulation pattern) 1
  Interventions: Device: Non-invasive brainstem stimulation
- Investigational Treatment 2 (Other): Investigational treatment mode (stimulation pattern) 2
  Interventions: Device: Non-invasive brainstem stimulation
- Investigational Treatment Mode - Open Label (Other): Investigational treatment mode (stimulation pattern)
  Interventions: Device: Non-invasive brainstem stimulation

INTERVENTIONS:
Device: Non-invasive brainstem stimulation — Study participants will self-administer ~19-minute treatments twice daily in the home setting over 24 weeks using a non-invasive brainstem modulation device. All participants will use the same treatment mode during the open label extension.

SUMMARY:
This is a double- blind, randomized controlled trial with an open label extension designed to evaluate the safety and potential efficacy of a non-invasive brainstem neuromodulation device for treating symptoms associated with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Up to 45 participants will first enter the double-blind, randomized controlled trial during which they will self-administer treatments twice daily in the home setting over 24 weeks with one of two investigational treatment modes. Participants who complete the randomized controlled trial will then enter the open label extension where all participants will self-administer twice-daily treatments over 24 weeks using the same investigational treatment mode that was reported to show benefit in a previous clinical trial in another neurodegenerative disease.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants (aged 65 - 85 years inclusive) diagnosed with probable Alzheimer's disease dementia .
* Willing and able to comply with study requirements.
* Have a study partner who sees the participant for more than three hours a day, 5x per week and is that is willing to consent and participate in the trial.
* Anticipation that the participant is able to remain on a stable regimen of medications used for the management of Alzheimer's disease and will not introduce new medications used to treat Alzheimer's disease during the study.
* Participant and study partner must both be fully vaccinated from COVID-19 prior to the study screen

Exclusion Criteria:

* Were diagnosed with probable Alzheimer's disease prior to 65 years of age.
* Has experienced a heart attack, angina, or stroke within the past 12 months or a transient ischemic attack (TIA) within the past 6 months.
* Are being treated with another neurostimulation device
* Experience frequent falls
* Works night shifts.
* Have unresolved complications from a previous surgical procedure at the baseline visit, such as swelling or persistent pain, that requires medical intervention.
* Have active ear infections, or other significant ear problems.
* Have a recent history of frequent ear infections
* Have a cochlear implant or hearing aids that cannot be easily/reliably removed for treatment.
* Have chronic tinnitus.
* Have previously been diagnosed with traumatic brain injury with ongoing sequela.
* History of medication-refractory depression or bipolar disorder in the past three years.
* History of schizophrenia.
* Participation in an interventional clinical trial for any medical or psychiatric indications within 3 months of the screening visit, or at any time during the study.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's Disease Assessment Scale-Cognitive-Plus (ADAS-Cog-14) | 24 weeks
  The ADAS-Cog-14 is a modified version of the Alzheimer's Disease Assessment Scale - Cognitive Subscale - a brief neuropsychological assessment developed to assess the level of cognitive dysfunction in AD. The scoring range is from 0 to 90, with higher scores indicating greater cognitive impairment.

SECONDARY OUTCOMES:
Change from baseline in the Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living (ADCS-iADL). | 24 weeks
  The ADCS-iADL is a 17-item subset of the Alzheimer's Disease Cooperative Study -Activities of Daily Living scale- an observer reported outcome that asks caregivers to rate the degree to which their family member or loved one can perform a variety of tasks. The scoring range is from 0 to 59 with higher scores indicated better performance.
Change from baseline in the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC). | 24 weeks
  The ADCS-CGIC is a clinician reported outcome that utilizes a systematic method for assessing clinically meaningful change taking input from both the participant and the informed other into account. The scale rates total change on a 7 point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse

OTHER OUTCOMES:
Change from baseline in The NeuroPsychiatric Inventory. | 24 weeks and 48 weeks
  a brief interview administered to caregivers to evaluate behavioral disturbances in dementia patients
Change from baseline in The Zarit Burden Interview. | 24 weeks and 48 weeks
  a measure of caregiver burden completed by caregivers
Change from baseline in The Mini- Mental State Exam. | 24 weeks and 48 weeks
  a widely used test of cognitive function among the elderly.
Change from baseline in the Alzheimer's Disease Cooperative Study -Activities of Daily Living. | 24 weeks and 48 weeks
  an observer reported outcome that asks caregivers to rate the degree to which their family member or loved one can perform a variety of tasks.
Change from baseline in the Symbol Digit Modality Test. | 24 weeks and 48 weeks
  a brief and commonly used test to evaluate processing speed.
Change from baseline in Phonemic Verbal Fluency Test. | 24 weeks and 48 weeks
  a brief measure of verbal functioning.
Change from baseline in the bloodborne biomarkers of neurodegeneration and blood-brain barrier permeability | 24 weeks and 48 weeks
  a biomarker for neurodegeneration
Change from baseline in the Alzheimer's Disease Assessment Scale-Cognitive-Plus (ADAS-Cog-14). | 48 weeks
  The ADAS-Cog-14 is a modified version of the Alzheimer's Disease Assessment Scale - Cognitive Subscale - a brief neuropsychological assessment developed to assess the level of cognitive dysfunction in AD. The scoring range is from 0 to 90, with higher scores indicating greater cognitive impairment.
Change from baseline in the Alzheimer's Disease Cooperative Study - instrumental Activities of Daily Living (ADCS-iADL). | 48 weeks
  The ADCS-iADL is a 17-item subset of the Alzheimer's Disease Cooperative Study -Activities of Daily Living scale- an observer reported outcome that asks caregivers to rate the degree to which their family member or loved one can perform a variety of tasks. The scoring range is from 0 to 59 with higher scores indicated better performance.
Change from baseline in the Alzheimer's Disease Cooperative Study - Clinical Global Impression of Change (ADCS-CGIC). | 48 weeks
  The ADCS-CGIC is a clinician reported outcome that utilizes a systematic method for assessing clinically meaningful change taking input from both the participant and the informed other into account. The scale rates total change on a 7 point scale:
  1. = Very much improved
  2. = Much improved
  3. = Minimally improved
  4. = No change
  5. = Minimally worse
  6. = Much worse
  7. = Very much worse

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Parkinson's Disease and Movement Disorders Center of Boca Raton, Boca Raton, Florida
  - USF Health Byrd Alzheimer's Institute, Tampa, Florida
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Riverside Neurology Specialists, Hampton, Virginia